CLINICAL TRIAL: NCT01515033
Title: Effect of Continuous and Interval Exercise Training on PETCO2 Response During Graded Exercise Test in Patients With Coronary Artery Disease
Brief Title: Aerobic Exercise on PETCO2 Response in Coronary Artery Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital TotalCor (Other)
Responsible Party: Principal Investigator, Danilo Marcelo Leite do Prado, MS, Hospital TotalCor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117/11
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Artery Disease; Exercise Addiction; Complication, Cardio-respiratory
Keywords: Coronary artery disease; Exercise; Ventilatory efficiency
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous exercise training (Experimental): The continuous exercise training was performed on a treadmill with a 50-minutes duration and intensity at ventilatory anaerobic threshold.
  Interventions: Other: aerobic exercise training
- interval exercise training (Experimental): The interval exercise training consisted of 7 sets of 3 minutes at respiratory compensation point and 7 sets of 3 minutes of exercise at moderate intensity corresponding to the ventilatory anaerobic threshold totaling 42 minutes
  Interventions: Other: aerobic exercise training

INTERVENTIONS:
Other: aerobic exercise training — The continuous exercise training was performed on a treadmill with a 50-minutes duration and intensity at ventilatory anaerobic threshold.
  The interval exercise training consisted of 7 sets of 3 minutes at respiratory compensation point and 7 sets of 3 minutes of exercise at moderate intensity corresponding to the ventilatory anaerobic threshold totaling 42 minutes
  Other Names: continuous training; interval training

SUMMARY:
The purpose of the present study was to evaluate: 1) the effects of continuous exercise training and interval exercise training on end-tidal carbon dioxide pressure (PETCO2) response during graded exercise test in patients with coronary artery disease; and 2) examine the effects of exercise training modalities on the association among PETCO2 at ventilatory anaerobic threshold (VAT) and indicators of ventilatory efficiency and cardiorespiratory fitness in patients with coronary artery disease.

DETAILED DESCRIPTION:
End-tidal carbon dioxide pressure (PETCO2) is a noninvasive index considered to be a good indicator in evaluating the ventilation/perfusion relationship in patients over a wide range conditions. Variations in PETCO2 have been shown to reflect changes in both cardiac output and pulmonary blood flow in animals and humans under constant ventilation. In this regard, it has been shown that patients with cardiac disease have an abnormally low PETCO2 during exercise, especially those with an impaired response of cardiac output during exercise

ELIGIBILITY:
Inclusion Criteria:

* was stable coronary artery disease diagnosed by coronary angiography

Exclusion Criteria:

* unstable angina pectoris,
* complex ventricular arrhythmias,
* pulmonary congestion and
* orthopaedic or neurological limitations to exercise

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-09; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
PetCO2 response during graded exercise test | before and after 3 months of the interventions
  End-tidal carbon dioxide pressure (PETCO2) is a noninvasive index considered to be a good indicator in evaluating the ventilation/perfusion relationship in patients over a wide range conditions (1,2). Variations in PETCO2 have been shown to reflect changes in both cardiac output and pulmonary blood flow in animals and humans under constant ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Danilo ML Prado, Prof.MS, Principal Investigator — Hospital TotalCor